CLINICAL TRIAL: NCT00521924
Title: Induction of Remission in RA Patients at Low Disease Activity by Additional Infliximab-therapy
Brief Title: Induction of Remission in RA Patients at Low Disease Activity by Additional Infliximab Therapy (Study P04644AM1) (TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: AESCA Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04644; 2005-004530-40
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Antirheumatic Agents; Methotrexate; Chloroquine; Leflunomide; Cyclosporine; Sulfasalazine; OM 89

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab + basic treatment (Experimental): 3 mg/kg infliximab plus basic treatment
  Interventions: Biological: infliximab
- Basic treatment (DMARDs) (Active Comparator): Rheumatoid Arthritis basic therapy (disease modifying anti-rheumatic drugs [DMARDs])
  Interventions: Drug: DMARDs (methotrexate; chloroquine; leflunomidum; cyclosporin A; sulfasalazine; OM 89.

INTERVENTIONS:
Biological: infliximab — infliximab 3 mg/kg and basic treatment
  Other Names: Basic treatment for RA (DMARDs)
  Arms: Infliximab + basic treatment
Drug: DMARDs (methotrexate; chloroquine; leflunomidum; cyclosporin A; sulfasalazine; OM 89. — Methotrexate (15 - 25 mg/week); chloroquine; leflunomidum; cyclosporin A; sulfasalazine; OM 89
  Arms: Basic treatment (DMARDs)

SUMMARY:
This Phase 3, randomized, open-label, multicenter study in rheumatoid arthritis (RA) patients with low disease activity (Disease Activity Score 28 [DAS28] >2.8 and <3.5) is being conducted to evaluate induction of remission by adding infliximab to pre-existing treatment versus no additional treatment. All subjects eligible for this study, aged >35 to <=65 years, will have a diagnosis of RA according to American College of Rheumatology (ACR) criteria, and will be offered additional treatment with infliximab. Prior to the start of treatment, subjects must be on a stable regimen of disease modifying antirheumatic drugs (DMARDs) for at least 3 months. Subjects will be randomized (1:1) to basic therapy with or without infliximab for a total duration of 38 weeks followed by a follow-up period of up to 6 months. Subjects randomized to basic therapy + infliximab will receive infliximab 3 mg/kg at Weeks 0, 2, 6, 14, 22, 30, and 38. The primary objective of the study is to assess the rate of remission according to DAS 28 (<2.6) at the end of treatment (after 38 weeks). Safety assessments include the incidence of adverse events, serious adverse events, and clinically notable abnormal vital signs and laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >35 and <=65 years with a diagnosis of rheumatoid arthritis (RA) according to American College of Rheumatology (ACR) criteria for at least 1 year and no more than 10 years prior to start of therapy; have active disease (Disease Activity Score [DAS] 28 >2.8 and <3.5), with changes in the DAS 28 score <0.6 within the 6 weeks before inclusion; have stable RA basic therapy according to standard criteria for at least 3 months; have a chest X-ray within 1 month prior to first infusion with no evidence of malignancy, infections, or fibrosis; and have screening laboratory test results that meet prespecified criteria. Patient must have at least one swollen joint. Patient must have evidence of erosive disease by x-ray at baseline.

Exclusion Criteria:

* Patients were excluded if they met any of the following criteria:

  * Women who are pregnant, nursing, or planning pregnancy within 15 months after screening (i.e., approximately 6 months following last infusion);
  * Use of any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer;
  * History of any other therapeutic agent targeted at reducing tumor necrosis factor (TNF);
  * History of previous administration of infliximab;
  * History of receiving human/murine recombinant products or has a known allergy to murine products;
  * Serious infection (such as hepatitis, pneumonia or pyelonephritis) in the previous 3 months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator.
  * Active tuberculosis (TB) or evidence of latent TB (positive purified protein derivative [PPD] skin test, a history of old or latent TB or chest X-ray without adequate therapy for TB initiated prior to first infusion of study drug), or evidence of an old or latent TB infection without documented adequate therapy. Patients with a current close contact with an individual with active TB and patients who have completed treatment for active TB within the previous 2 years are explicitly excluded from the trial. Patients with a household member who has a history of active pulmonary TB should have had a thorough evaluation for TB prior to study enrollment as recommended by a local infectious disease specialist or published local guidelines of TB control agencies.
  * Hepatitis B surface antigen or Hepatitis C (HCV) antibody positive; documented Human Immunodeficiency Virus (HIV) infection;
  * Have an opportunistic infection, including but not limited to evidence of active cytomegalovirus, active pneumocystis carinii, aspergillosis, or atypical mycobacterium infection, etc, within the previous 6 months;
  * Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, psychiatric, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis);
  * Concomitant congestive heart failure >= New York Heart Association (NYHA) II;
  * Have a transplanted organ (with the exception of a corneal transplant >3 months prior to screening);
  * Fibromyalgia;
  * Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence);
  * History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy of unusual size or location (such as nodes in the posterior triangle of the neck, infraclavicular, epitrochlear, or peri-aortic areas), or splenomegaly; or
  * Known recent substance abuse (drug or alcohol).

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to poor enrollment rate, this trial was terminated prematurely. Eight patients had been enrolled from June 2007 to April 2008: 4 in each arm.
Period: Overall Study
Arm/Group | Infliximab + Basic Treatment | Basic Treatment (DMARDs)
Started | 4 (Subjects randomized) | 4 (Subjects randomized)
Completed | 0 (At Early Termination, 1 patient completed Week 2 and 2 patients completed Week 6.) | 0 (At Early Termination, 3 patients completed Week 6 and 1 completed Week 22.)
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab + Basic Treatment | Basic Treatment (DMARDs) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Customized [Number; unit: participants] | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Remission According to Disease Activity Score (DAS) 28 (< 2.6)
Description: The DAS 28 is an assessment of disease activity based on swollen joint count, erythrocyte sedimentation rate, and general health. Patients can be scored on a range of 0 to 10, with lower scores indicating less disease activity.
Time Frame: after 38 weeks
Population: This trial terminated early due to poor enrollment. Since none of the randomized patients reached Week 38, no change of DAS28 between baseline and Week 38 could be analyzed.
Arm/Group | Infliximab + Basic Treatment | Basic Treatment (DMARDs)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: DAS 28 at Baseline vs at Week 38; Quality of Life; American College of Rheumatology (ACR) Response Disease Progression (X-ray); Effect of Inflammatory Markers on Response and Disease Progression; Assess Simplified Disease Activity Index (SDAI).
Description: These were not prespecified key secondary outcomes; therefore, results will not be disclosed.
Time Frame: Weeks 14, 38, and 62
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Infliximab + Basic Treatment | Basic Treatment (DMARDs)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) has the right to publish/publicly present the results of the Study, but may not to publish/publicly present any interim results. PI must provide 45 days written notice to Sponsor prior to submission for publication/presentation to permit Sponsor to review drafts for publication which report any results arising out of the Study. Sponsor shall have the right to review and comment on any Public Presentation.